CLINICAL TRIAL: NCT01514214
Title: A Randomized Trial Comparing a Winged Perimeter Stent and Traditional Polyethylene Plastic Stent in the Management of Malignant Distal Biliary Strictures
Brief Title: Winged Perimeter Versus Traditional Plastic Biliary Stent for Malignant Bile Duct Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Telford, Clinical Professor of Medicine, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H10-02829
Record Dates: First submitted 2012-01-16; First posted 2012-01-23 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Malignant Tumor of Extrahepatic Bile Duct
Keywords: ERCP; biliary stricture; viaduct; cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Winged perimeter stent (Active Comparator): Patients who receive the Viaduct stent during ERCP
  Interventions: Device: WInged perimeter biliary stent insertion (Viaduct)
- polyethylene stent arm (Active Comparator): Patient who receive the traditional polyethylene stent during ERCP
  Interventions: Device: traditional polyethylene stent insertion (Cotton Huibregtse)

INTERVENTIONS:
Device: WInged perimeter biliary stent insertion (Viaduct) — Insertion of a winged perimeter stent. Size to be determined during the ERCP based on findings.
  Other Names: Viaduct Stent
  Arms: Winged perimeter stent
Device: traditional polyethylene stent insertion (Cotton Huibregtse) — insertion of a traditional polyethylene stent during ERCP, size to be determined depending on findings during ERCP
  Other Names: Cotton Huibregtse Stent
  Arms: polyethylene stent arm

SUMMARY:
Strictures in the bile duct cause a blockage of flow of bile. This leads to potential problems including jaundice, itch and infection in the bile duct. The usual first step in this situation would be to allow flow of bile by placing a stent across the stricture. This is usually done by a special type of endoscopy procedure called an endoscopic retrograde cholangiopancreatography, or ERCP.

The most commonly used stent are made from a plastic material called polyethylene and has a central lumen in which bile drains through it. Health Canada has approved the sale and use of another stent with a winged perimeter (the VIADUCT stent) for placement in bile duct strictures and is used routinely in our hospitals. However, the investigators do not know which stent is better at treating bile duct strictures. In order to determine which stent would be more useful, the VIADUCT stent and the usual polyethylene flanged stent must be studied under carefully controlled circumstances. This will be done by a randomized, subject-blinded study. Other trials in the past have looked at other stents in this way, but this is the first time the VIADUCT stent has been looked at in this manner. The investigators suspect that the design of the VIADUCT stent will allow it to work for a longer period of time compared to the traditional polyethylene stent.

DETAILED DESCRIPTION:
Biliary obstruction usually presents with jaundice, pruritis, cholangitis, and steatorrhoea. Strictures which are a common cause of biliary obstruction, may be secondary to benign or malignant conditions. Common benign conditions include chronic pancreatitis, primary sclerosing cholangitis, autoimmune pancreatitis, prior surgery and recurrent pyogenic cholangitis. Cholangiocarcinomas, ampullary and pancreatic tumours are more common causes of malignant biliary obstruction.

The principles of managing biliary strictures are to determine the underlying cause of the stricture, whilst achieving drainage of the biliary tree, initially with the placement of a plastic stent via an endoscopic retrograde cholangiopancreatography (ERCP). Strictures are sampled using biliary brush cytology and/or biliary biopsy to assess for underlying malignancy. Malignant strictures are usually staged for resectability with computed tomography (CT), magnetic resonance cholangiopancreatography (MRCP) and/or endoscopic ultrasound (EUS).

The Viaduct stent (GI Supply, Camp Hill, Pennsylvania, USA) is a unique stent design and has a winged perimeter, which channels flow of bile around the stent, rather than through a central lumen. Theoretically this may enhance flow and biliary drainage, and prevent obstruction. Both polyethylene and Viaduct plastic stents are approved for use by Health Canada for benign and malignant biliary conditions. It is not known whether one stent is superior to the other in maintaining symptomatic relief from bile duct strictures as there have been no studies to date comparing the two stents.

There is limited published data on the Viaduct stent. A pilot study of the winged stent design was published in 2006. Five patients had winged stents inserted and followed for 2 weeks. The were no problems with stent insertion and symptoms of obstruction and jaundice improved over this time. One study published in abstract form retrospectively compared 34 Viaduct stents matched with 240 "conventional" stents over a five year period. There was no statistical difference with stent dysfunction, and a trend towards patency with the Viaduct stent.

The primary aim of this study is to compare the stent patency time in the Viaduct and polyethylene stent groups in subjects with malignant bile duct strictures. The secondary aims are to determine the etiology of stent failure in the two treatment groups, to identify and compare device-related adverse events in the two treatment groups, to identify other patient factors associated with stent failure, and to compare survival between the Viaduct and polyethylene stent groups.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Bile duct stricture confirmed on cholangiography at ERCP
* Malignant etiology confirmed on histology or cytology
* Duct stricture is > 1 cm distal to the biliary hilum (bifurcation of the common hepatic duct into the right and left hepatic ducts)

Exclusion Criteria:

* Unable to obtain consent
* Unable to tolerate procedure
* Hilar strictures
* Known benign biliary strictures and benign strictures confirmed after randomization
* Circumstances where an alternative biliary stent (pigtail stent or metal stent) is deemed critical by the treating Gastroenterologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Stent patency time | six months post stent insertion
  Time to bile duct re-obstruction

SECONDARY OUTCOMES:
Etiology of stent failure | six months post stent insertion
  Usually occlusion or migration
Compare number of patients with device related adverse events | six months post stent insertion
  Comparing both procedural and delayed complications of stents
Identify patient factors associated with stent failure | six months post stent insertion
Survival between the two groups | six months post stent insertion
  Measurement in months of survival post diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Telford, MD MPH FRCPC, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raju GS, Sud R, Elfert AA, Enaba M, Kalloo A, Pasricha PJ. Biliary drainage by using stents without a central lumen: a pilot study. Gastrointest Endosc. 2006 Feb;63(2):317-20. doi: 10.1016/j.gie.2005.07.053. PMID 16427942